CLINICAL TRIAL: NCT04277624
Title: A Phase 1 Crossover Study to Assess the Bioequivalence of Fezolinetant Following a Single Dose of Fezolinetant (Test Formulation) Compared to a Single Dose of Fezolinetant Phase 3 Formulation (Reference Formulation) in Healthy Female Subjects
Brief Title: A Study to Assess Bioequivalence of Fezolinetant Formulations in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2693-CL-0010
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: fezolinetant; ESN364; menopause
MeSH Terms: interventions — fezolinetant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fezolinetant: Test Formulation then Reference Formulation (Experimental): Participants will receive a single oral dose of fezolinetant test formulation on day 1 of study period 1. After a washout of 5 days the participants will receive a single oral dose of fezolinetant reference formulation on day 1 of study period 2.
  Interventions: Drug: fezolinetant - test formulation; Drug: fezolinetant - reference formulation
- Fezolinetant: Reference Formulation then Test Formulation (Experimental): Participants will receive a single oral dose of fezolinetant reference formulation on day 1 of study period 1. After a washout of 5 days the participants will receive a single oral dose of fezolinetant test formulation on day 1 of study period 2.
  Interventions: Drug: fezolinetant - test formulation; Drug: fezolinetant - reference formulation

INTERVENTIONS:
Drug: fezolinetant - test formulation — Administered orally
  Other Names: ESN364
Drug: fezolinetant - reference formulation — Administered orally
  Other Names: ESN364

SUMMARY:
The purpose of this study is to assess the bioequivalence of a single dose of fezolinetant test formulation compared to a single dose of fezolinetant reference formulation under fasting conditions. This study will also evaluate the safety and tolerability of a single dose of fezolinetant test formulation and a single dose of fezolinetant reference formulation.

DETAILED DESCRIPTION:
Each participant will participate in 2 study periods separated by a washout of at least 5 days between investigational product (IP) administrations. Participants will be randomized to 1 of 2 sequences: either fezolinetant test formulation followed by fezolinetant reference formulation or fezolinetant reference formulation followed by fezolinetant test formulation. Participants will be admitted to the clinical unit on day -1 and will be residential for 2 study periods for a total of 10 days/9 nights. Premenopausal female participants will be admitted to the clinical unit during days 1 to 3 of their menstrual cycle. Participants will receive a single dose of test formulation or reference formulation under fasting conditions on day 1 of each period i.e., days 2 to 4 (period 1) and days 7 to 9 (period 2) of their menstrual cycle for premenopausal female participants. Participants are to remain semirecumbent and avoid lying on either the left or right side for 4 hours postdose. Pharmacokinetic samples will be collected predose on day 1 of each period and at multiple time points postdose. Standard safety and tolerability assessments will be conducted. Participants will be discharged from the clinical unit on day 4 of period 2 on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit.

The study will be completed with an end-of-study visit (ESV). The ESV will take place 5 to 9 days after discharge from period 2 or at early discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy female subject.
* Subject has a body mass index (BMI) range of 18.5 to 34.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Postmenopausal female subjects only: Subject is postmenopausal according to 1 of the following criteria:

  * Spontaneous amenorrhea for ≥ 12 consecutive months
  * Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] > 40 IU/L); or
  * Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit (with or without hysterectomy)
* Subject agrees not to participate in another interventional study while participating in the present study.
* Premenopausal female subjects only: Subject has had a regular menstrual cycle (from 25 to 31 days ± 3 days) for 3 months prior to starting the IP administration.
* Premenopausal female subjects only: Subject is not pregnant and at least meets 1 of the following criteria:

  * If the subject is not of childbearing potential: Subject has lost fertility permanently by surgery excluding oophorectomy (e.g., hysterectomy, bilateral salpingectomy).
  * If the subject is a woman of childbearing potential (WOCBP): Subject agrees to follow the contraceptive guidance from the time of providing informed consent through at least 30 days after the final IP administration. However, if the subject's partner has lost fertility by surgery (vasectomy or bilateral orchiectomy) etc., confirmed with documentation of both the procedure and absence of sperm, it is not necessary to implement contraceptive methods.

Note: If absence of sperm cannot be confirmed in the subject's partner who received a vasectomy, an alternative contraceptive method must be used.

* Premenopausal female subjects only: Subject agrees not to breastfeed or donate ova from the time of providing informed consent until 30 days after the last IP administration.

Exclusion Criteria:

* Subject has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has a known or suspected hypersensitivity to fezolinetant or any components of the formulations used.
* Subject has had previous exposure with fezolinetant.
* Subject has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) > 1.5 × upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first investigational product (IP) administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 45 or > 90 bpm or hypertension as defined by a systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 80 mmHg based on the average of 3 readings on at least 2 different occasions during the screening period.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) of > 470 msec on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, contraception [oral, injectable, implantable or transdermal] and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first IP administration and for hormone replacement therapy (HRT) in the 8 weeks prior to first IP administration, except for occasional use of acetaminophen (up to 2 g/day) and topical dermatological products, including corticosteroid products.
* Subject has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening.
* Subject has a history of consuming > 7 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol at screening or on day -1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the subject tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Subject has used any inducer of cytochrome P450 (CYP) 1A2 in the 3 months prior or inhibitors of CYP 1A2 in the 2 weeks or 5 half-lives of the inhibitor, whichever is longer, prior to day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B core antibodies, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.
* Premenopausal female subjects only: Subject has been pregnant within 6 months or has been breastfeeding within 3 months prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of fezolinetant in plasma: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 72 hours postdose in each study period
  AUCinf will be recorded from the pharmacokinetic (PK) plasma samples collected
Pharmacokinetics (PK) of fezolinetant in plasma: Area under the concentration-time curve (AUC) from the time of dosing to the last measurable concentration (AUClast) | Up to 72 hours postdose in each study period
  AUClast will be recorded from the pharmacokinetic (PK) plasma samples collected
Pharmacokinetics (PK) of fezolinetant in plasma: Maximum concentration (Cmax) | Up to 72 hours postdose in each study period
  Cmax will be recorded from the pharmacokinetic (PK) plasma samples collected

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 19 days
  An AE is any untoward medical occurrence in a subject administered an investigatonal product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 19 days
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 19 days
  Number of participants with potentially clinically significant vital sign values.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- PAREXEL Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.